CLINICAL TRIAL: NCT03082716
Title: Custodiol Versus Blood Cardioplegaia in Paediatric Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB 2016-08 Custodiol Study
Record Dates: First submitted 2017-01-29; First posted 2017-03-17 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Congenital Heart Disease
Keywords: cardioplegia; myocardial protection; custodiol; htk
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Bretschneider cardioplegic solution; Receptor, EphB4

STUDY DESIGN:
Intervention Model Description: Randomisation :
  Computer generated randomisation into two groups based on cardioplegia solution .
  if randomised to blood patient will receive blood cardioplegia, delivered by microplegia delivery system by adding potassium to the blood (K= 35 ml eq/L) . The initial dose will be 35ml/ kg, and subsequent doses 20-15 ml/kg given every 20 minutes at a Temperature of 10 - 15 °C, while maintaining a perfusion pressure of 100-125 mmHg.
  if randomised to custodial patient will receive single dose of HTK custodiol cardioplegia. at temperature of 4-8°C and will be perfused for 6-8 minutes. Dose will start from 400 up to 1000 ml according to the child's body weight. Perfusion pressure will be kept at 70 - 80 mmHg until the heart is arrested.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding :
  Surgeons will know the type of cardioplegia in the OR while other assessor will be blinded .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- blood cardioplegia group (Active Comparator): patient will receive blood cardioplegia, delivered by microplegia delivery system by adding potassium to the blood (K= 35 ml eq/L) . The initial dose will be 35ml/ kg, and subsequent doses 20-15 ml/kg given every 20 minutes at a Temperature of 10 - 15 °C, while maintaining a perfusion pressure of 100-125 mmHg.
  Interventions: Drug: Blood cardioplegia
- custodiol group (Experimental): patient will receive single dose of HTK custodiol cardioplegia. at temperature of 4-8°C and will be perfused for 6-8 minutes. Dose will start from 400 up to 1000 ml according to the child's body weight. Perfusion pressure will be kept at 70 - 80 mmHg until the heart is arrested.
  Interventions: Drug: Custodiol Solution

INTERVENTIONS:
Drug: Custodiol Solution — After cross clamping patient will receive single dose of HTK custodiol cardioplegia. at temperature of 4-8°C and will be perfused for 6-8 minutes. Dose will start from 400 up to 1000 ml according to the child's body weight. Perfusion pressure will be kept at 70 - 80 mmHg until the heart is arrested.
  Other Names: htk
  Arms: custodiol group
Drug: Blood cardioplegia — After cross clamping patient will receive blood cardioplegia, delivered by microplegia delivery system by adding potassium to the blood (K= 35 ml eq/L) . The initial dose will be 35ml/ kg, and subsequent doses 20-15 ml/kg given every 20 minutes at a Temperature of 10 - 15 °C, while maintaining a perfusion pressure of 100-125 mmHg.
  Arms: blood cardioplegia group

SUMMARY:
Cardioplegic arrest is an essential part of cardiac surgery which aims to allow myocardial preservation and minimise myocardial swelling ,while providing a motionless and bloodless field ,.Blood cardioplegia has proven its efficacy for several decades and surgeons are still preferring to use it for myocardial protection of paediatric cardiac surgery ,although it is thought to be more time consuming since it is given with interrupted doses, . Even when advancement has came along the field of myocardial protection and cardioplegia solutions with the introduction of Bretschneider Histidine-Tryptophan-Ketoglutarate solution ,custodiol ,in 1970 ,which is given as a single dose and believed to be convenient, simple to deliver , and less time consuming . Many Surgeons haven't change their practice possibly due to paucity of studies comparing cardioplegia solutions in paediatric cardiac surgery and conflicting reports regarding the superiority of different cardioplegia solution.The investigators aim to provide evidence that will help paediatric cardiac surgeons to choose the optimal solution for their practice .

DETAILED DESCRIPTION:
Hypothesis :

Custodial is not inferior to blood cardioplegia in myocardial protection in paediatric cardiac surgery ..

Methodology :

Study design :

Randomized controlled trial

Data collection:

All demographic data ,diagnosis ,procedure(type.CPB time ,crossclamp time) , surgeon and hospital course details .

Computer generated randomisation into two groups based on cardioplegia solution .

if randomised to blood patient will receive blood cardioplegia, delivered by microplegia delivery system by adding potassium to the blood (K= 35 ml eq/L) . The initial dose will be 35ml/ kg, and subsequent doses 20-15 ml/kg given every 20 minutes at a Temperature of 10 - 15 °C, while maintaining a perfusion pressure of 100-125 mmHg.

if randomised to custodial patient will receive single dose of HTK custodiol cardioplegia. at temperature of 4-8°C and will be perfused for 6-8 minutes. Dose will start from 400 up to 1000 ml according to the child's body weight. Perfusion pressure will be kept at 70 - 80 mmHg until the heart is arrested..

Blinding :

Surgeons will know the type of cardioplegia in the OR while other assessor will be blinded .

Sample size calculated with an online calculator based on α error of 0.05 and β error of 0.2 to detect an absolute risk difference of 15% in composite end point between the two groups yielded 137 in each arm ,The results will be presented as mean (SD), median (interquartile range), or proportion . Using relative risk and log rank for statistical analysis .A P value of less than 0.05 will be considered statistically significant. Statistical analyses will be carried out using the SPSS .

Safety monitoring and interim results :

Both cardioplegia solutions are already in use and FDA approved there is no safety concerns at the time being . However , an interim analysis will be carried on every 6 months and the principal investigator will decide weather to stop or carry on if any major discrepancies in outcomes

literature review : After an extensive literature review the investigators found only one randomised trial by elmorsy et al , which concluded that A single dose of an HTK cardioplegic solution provides better myocardial and cerebral protection than repeated doses of oxygenated blood cardioplegia during pediatric congenital cardiac surgery.

On the other hand there was another retrospective report by bojan et al, found that The use of Custodiol cardioplegia in neonates undergoing ASO was associated with a larger troponin release when compared with warm blood cardioplegia,p <0.001 suggesting poor myocardial protection.

koruon et al, done a tissue level comparison between htk and conventional crystalloid cardioplegia and their statistical analysis revealed no significant difference between the two groups regarding the clinical variables, apoptotic indices and proliferation indices.

Liu j et al ,did a retrospective study comparing custodiol to St. Thomas crystalloid cardioplegia which concluded That HTK group had shorter cross-clamping time and more frequent spontaneous defibrillation than St. Thomas group.

Also an animal study by Chen Y et al, on piglets that were randomised to either a single dose of HTK or multidose cold blood cardioplegia .. No significant differences were noted in the myocardial lactate content, ATP content, and histopathological score between both groups .

Finally a retrospective report by E Qulisy et al concluded that Custodiol cardioplegia is associated with less myocardial protection and higher adverse outcomes compared to blood cardioplegia in pediatric age group undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* All paediatric patients referred to our hospital which will undergo open cardiac repair with cardiopulmonary bypass and cardioplegic arrest .

Exclusion Criteria:

* All emergency procedure( require immediate surgery)
* Cases that don't require use of cardioplegia .

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Mortality (yes/no) | up to 30 days
  Death of all causes
ICU stay (days) | up to 90 days (length of ICU stay required after the operative procedure recorded by days until discharge or death)
  length of ICU stay
Arrhythmia (yes/no) | up to 48 hours
  post operative arrythmia that required intervention

SECONDARY OUTCOMES:
length of stay (days) | up to 90 days (length of the hospital stay required since admission recorded by days until discharge or death )
length of mechanical ventilation (hours) | up to 5 days
myocardial biomarkers | up to 5 days
  (troponin and CKMB) measured (preoperatively,postoperatively 6h,24h,48h,)
Subjective ventricular function (normal,mildly depressed ,moderately depressed ,moderately-severe depressed ,severly depressed ) | up to 24 hours
  assessed by a cardiologist subjective assessment of the echocardiographically (preoperative ,immediate post repair ,24h post operative )
Ejection fraction (percentage) | up to 24 hours
  assessed by echocardiography (preoperative ,immediate post repair ,24h post operative )
ECMO support (yes/no) | intraoperative
vasoactive inotropic score ( low or high) | up to 48 hour
  Vasoactive Inotropic score : (all doses of inotropes recorded hourly during 48 h)
  Dopamine dose (μg/kg/min) + Dobutamine dose (μg/kg/min) +100 × epinephrine dose (μg/kg/min)+ 10 X Milrinone dose (μg/kg/min) +10,000 × Vasopressin dose (U/kg/min) + 100 × Norepinephrine dose (μg/kg/min)
  calculated hourly for 48 hours and added than divided by 48 to give the score . if maximum score < 20 its low VIS and if maximum score ≥ 20 its a high VIS

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Centre, Jeddah, Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kotani Y, Tweddell J, Gruber P, Pizarro C, Austin EH 3rd, Woods RK, Gruenwald C, Caldarone CA. Current cardioplegia practice in pediatric cardiac surgery: a North American multiinstitutional survey. Ann Thorac Surg. 2013 Sep;96(3):923-9. doi: 10.1016/j.athoracsur.2013.05.052. Epub 2013 Jul 31. PMID 23915588
- [Background] Harvey B, Shann KG, Fitzgerald D, Mejak B, Likosky DS, Puis L, Baker RA, Groom RC; American Society of ExtraCorporeal Technology's International Consortium for Evidence-Based Perfusion and Pediatric Perfusion Committee. International pediatric perfusion practice: 2011 survey results. J Extra Corpor Technol. 2012 Dec;44(4):186-93. PMID 23441558
- [Background] Korun O, Ozkan M, Terzi A, Askin G, Sezgin A, Aslamaci S. The comparison of the effects of Bretschneider's histidine-tryptophan-ketoglutarate and conventional crystalloid cardioplegia on pediatric myocardium at tissue level. Artif Organs. 2013 Jan;37(1):76-81. doi: 10.1111/j.1525-1594.2012.01575.x. PMID 23305576
- [Background] elmorsy et al , Does type of cardioplegia affect myocardial and cerebral outcome in pediatric open cardiac surgeries? Ain-Shams Journal of Anesthesiology ,2014; 2(7) :242-249
- [Result] Bojan M, Peperstraete H, Lilot M, Tourneur L, Vouhe P, Pouard P. Cold histidine-tryptophan-ketoglutarate solution and repeated oxygenated warm blood cardioplegia in neonates with arterial switch operation. Ann Thorac Surg. 2013 Apr;95(4):1390-6. doi: 10.1016/j.athoracsur.2012.12.025. Epub 2013 Feb 22. PMID 23462260
- [Result] Liu J, Feng Z, Zhao J, Li B, Long C. The myocardial protection of HTK cardioplegic solution on the long-term ischemic period in pediatric heart surgery. ASAIO J. 2008 Sep-Oct;54(5):470-3. doi: 10.1097/MAT.0b013e318188b86c. PMID 18812735
- [Result] Chen Y, Liu J, Li S, Li W, Yan F, Sun P, Wang H, Long C. Which is the better option during neonatal cardiopulmonary bypass: HTK solution or cold blood cardioplegia? ASAIO J. 2013 Jan-Feb;59(1):69-74. doi: 10.1097/MAT.0b013e3182798524. PMID 23263337
- [Result] Custodiol versus blood cardioplegia in pediatric cardiac surgery. SHAJ .October 2015 ;27,(4):327
- [Derived] Elmahrouk AF, Shihata MS, Al-Radi OO, Arafat AA, Altowaity M, Alshaikh BA, Galal MN, Bogis AA, Al Omar HY, Assiri WJ, Jamjoom AA. Custodiol versus blood cardioplegia in pediatric cardiac surgery: a randomized controlled trial. Eur J Med Res. 2023 Oct 5;28(1):404. doi: 10.1186/s40001-023-01372-4. PMID 37798628